CLINICAL TRIAL: NCT00005945
Title: Escalating Dose Intravenous Methotrexate Without Leucovorin Rescue Versus Oral Methotrexate and Single Versus Double Delayed Intensification for Children With Standard Risk Acute Lymphoblastic Leukemia
Brief Title: Comparison of Different Combination Chemotherapy Regimens in Treating Children With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1991; CCG-1991 (Other: Children's Cancer Group); CDR0000067855 (Other: Clinical Trials.gov); NCT00005945 (Other: NCI); NCI-2012-02333 (Other: NCI); U10CA098543 (NIH)
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia; L1 childhood acute lymphoblastic leukemia; L2 childhood acute lymphoblastic leukemia; L3 childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; Doxorubicin; Mercaptopurine; Methotrexate; pegaspargase; Thioguanine; Vincristine; Radiotherapy; Radiation; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Induction Not Randomized (Experimental): Standard Induction (28 Days). M3 Marrow at Day 28 and Off Protocol Therapy.
  Interventions: Drug: cyclophosphamide; Drug: dexamethasone; Drug: methotrexate; Drug: pegaspargase; Drug: vincristine sulfate
- Induction and Oral MTX, Double Delayed Intensification CNS (Experimental): Patients with CNS disease at diagnosis, without other unfavorable characteristics. Standard Induction (28 Days). Consolidation (28 days) and in remission Day 21 and at time of randomization, Interim maintenance I (2 months), Delayed intensification I (2 months), Interim maintenance II (2 months), Delayed intensification II (2 months), then Maintenance (12 week cycles). Cranial radiation therapy during the Consolidation phase.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy
- Induction and Augmented regimen (IV MTX, Double DI) (Experimental): Patients with unfavorable characteristics. Standard Induction (14 Days), Augmented Induction (Days 14-35), Consolidation (9 weeks), Interim Maintenance I (56 Days), Delayed Intensification I (2 months), Interim Maintenance II (2 months), Delayed Intensification II (2 months), then Maintenance (84 day courses).
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy
- Induction and Oral MTX, Single Delayed Intensification (Experimental): Patients without CNS disease at diagnosis, with favorable cytogenetics. Standard Induction (28 Days). Consolidation (28 days) and in remission Day 21 and at time of randomization, Interim maintenance I (2 months), Delayed intensification I (2 months), Interim maintenance II (2 months) then Maintenance (12 week cycles). Biopsy-proven testicular leukemia pts at diagnosis will receive testicular radiation therapy during the consolidation phase.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy
- Induction and Oral MTX, Double Delayed Intensification (Experimental): Patients without CNS disease at diagnosis, with favorable cytogenetics. Standard Induction (28 Days). Consolidation (28 days) and in remission Day 21 and at time of randomization, Interim maintenance I (2 months), Delayed intensification I (2 months), Interim maintenance II (2 months), Delayed intensification II (2 months), then Maintenance (12 week cycles). Biopsy-proven testicular leukemia pts at diagnosis will receive testicular radiation therapy during the consolidation phase.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy
- Induction and IV MTX, Single Delayed Intensification (Experimental): Patients without CNS disease at diagnosis, with favorable cytogenetics. Standard Induction (28 Days). Consolidation (28 days) and in remission Day 21 and at time of randomization, Interim maintenance I (2 months), Delayed intensification I (2 months), Interim maintenance II (2 months) then Maintenance (12 week cycles). Biopsy-proven testicular leukemia pts at diagnosis will receive testicular radiation therapy during the consolidation phase.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy
- Induction and IV MTX, Double Delayed Intensification (Experimental): Patients without CNS disease at diagnosis, with favorable cytogenetics. Standard Induction (28 Days). Consolidation (28 days) and in event free remission Day 21 and at time of randomization, Interim maintenance I (2 months), Delayed intensification I (2 months), Interim maintenance II (2 months), Delayed intensification II (2 months), then Maintenance (12 week cycles). Biopsy-proven testicular leukemia pts at diagnosis will receive testicular radiation therapy during the consolidation phase.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxan; NSC-26271
Drug: cytarabine — Given IT
  Other Names: Cytosine Arabinoside; Ara_C; Cytosar-U; NSC-63878
  Arms: Induction and Augmented regimen (IV MTX, Double DI); Induction and IV MTX, Double Delayed Intensification; Induction and IV MTX, Single Delayed Intensification; Induction and Oral MTX, Double Delayed Intensification; Induction and Oral MTX, Double Delayed Intensification CNS; Induction and Oral MTX, Single Delayed Intensification
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Cerubidine; NSC-82151
  Arms: Induction and Augmented regimen (IV MTX, Double DI)
Drug: dexamethasone — Given PO
  Other Names: Decadron; DM; NSC-34521
Drug: doxorubicin hydrochloride — Dose 25 g/m² IV Days 0, 7, 14, given over a period of 15 minutes to 2 hours
  Other Names: Adriamycin; NSC-123127
  Arms: Induction and Augmented regimen (IV MTX, Double DI); Induction and IV MTX, Double Delayed Intensification; Induction and IV MTX, Single Delayed Intensification; Induction and Oral MTX, Double Delayed Intensification; Induction and Oral MTX, Double Delayed Intensification CNS; Induction and Oral MTX, Single Delayed Intensification
Drug: mercaptopurine — Given PO
  Other Names: 6-MP
  Arms: Induction and Augmented regimen (IV MTX, Double DI); Induction and IV MTX, Double Delayed Intensification; Induction and IV MTX, Single Delayed Intensification; Induction and Oral MTX, Double Delayed Intensification; Induction and Oral MTX, Double Delayed Intensification CNS; Induction and Oral MTX, Single Delayed Intensification
Drug: methotrexate — Given PO and IT
  Other Names: MTX
Drug: pegaspargase — Given IM
  Other Names: PEG-asparaginase; Oncaspar; L-asparaginase with polyethylene glycol
Drug: thioguanine — Given PO
  Other Names: 6 TG; NSC-752
  Arms: Induction and Augmented regimen (IV MTX, Double DI); Induction and IV MTX, Double Delayed Intensification; Induction and IV MTX, Single Delayed Intensification; Induction and Oral MTX, Double Delayed Intensification; Induction and Oral MTX, Double Delayed Intensification CNS; Induction and Oral MTX, Single Delayed Intensification
Drug: vincristine sulfate — Given IV
  Other Names: Oncovin; NSC-67574; VCR
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy; radiation
  Arms: Induction and Augmented regimen (IV MTX, Double DI); Induction and IV MTX, Double Delayed Intensification; Induction and IV MTX, Single Delayed Intensification; Induction and Oral MTX, Double Delayed Intensification; Induction and Oral MTX, Double Delayed Intensification CNS; Induction and Oral MTX, Single Delayed Intensification

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Giving more than one drug may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating childhood acute lymphoblastic leukemia.

PURPOSE: This randomized phase III trial is comparing different combination chemotherapy regimens to see how well they work in treating children with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the event-free survival and overall survival of children with standard-risk acute lymphoblastic leukemia treated with escalating-dose IV methotrexate without leucovorin calcium versus oral methotrexate during the interim maintenance phase of therapy.
* Compare the event-free survival and overall survival of these patients after receiving treatment in two delayed intensification phases versus one delayed intensification phase.
* Compare the toxic effects of oral versus escalating-dose intravenous methotrexate in these patients.
* Determine the prognostic significance of the rate of disappearance of peripheral lymphoblasts and lymphocytes during the first week of treatment in these patients.
* Determine the prognostic significance of trisomies of chromosomes 4, 5, 10, and 17 and early treatment response in patients treated with these regimens.
* Determine the prognostic significance of the TEL-AML1 fusion transcript and early treatment response in patients treated with these regimens.
* Determine the minimal residual disease (MRD) by polymerase chain reaction in bone marrow and cerebrospinal fluid at various stages of therapy in these patients.
* Determine the prognostic significance of MRD during various stages of therapy in these patients.
* Determine whether a second delayed intensification therapy improves the prognosis of patients who have MRD at the end of induction therapy.

OUTLINE: This is a randomized, multicenter study. Patients without CNS disease at diagnosis, achieving a specified early marrow response profile and M1 marrow status of less than 5% blasts in the bone marrow (regardless of the proportion of mature lymphocytes) by day 28 of induction therapy, and remaining event free with favorable bone marrow status and cytogenetics between day 21 and 28 of consolidation therapy are randomized to one of four treatment arms. Patients with CNS disease at diagnosis are assigned to treatment arm II and undergo cranial irradiation. Patients with any of the following unfavorable bone marrow features and/or unfavorable cytogenetic features are assigned to the augmented treatment regimen by day 21 of induction chemotherapy or at the beginning of consolidation chemotherapy:

NOTE: All T-cell precursor patients that are not more than 4 months past completion of the delayed intensification phase of therapy should be switched to the augmented regimen as of 3/8/2004. These patients may be switched to the augmented regimen. The protocol gives specific instructions according to the phase of therapy the patients are actually in.

* Unfavorable marrow status:

  * M2: 5-25% blasts in bone marrow at day 28 of induction chemotherapy (or at day 14 of induction chemotherapy if day 7 status is M3) OR
  * M3: More than 25% blast cell in bone marrow, regardless of the proportion of mature lymphocytes at day 14 of induction chemotherapy
* Unfavorable cytogenetics: Must have 1 of the following:

  * t(9;22)(q34;q11)
  * t(4;11)(q21;q23)
  * Balanced t(1;19)(q23;p13)
  * Hypodiploidy with less than 45 chromosomes
  * Other 11q23 translocations involving MLL Patients receive standard induction chemotherapy comprising cytarabine (ARA-C) intrathecally (IT) on day 0 or up to 72 hours before day 0; oral dexamethasone (DM) twice daily on days 0-27; vincristine (VCR) IV on days 0, 7, 14, and 21; and pegaspargase (PEG-ASP) intramuscularly (IM) once between days 3-5. Patients without CNS disease at diagnosis receive methotrexate (MTX) IT on days 7 and 28. Patients with CNS disease at diagnosis receive MTX IT on days 7, 14, 21, and 28.

Patients who have achieved M1 marrow status by day 28 of induction therapy and have favorable early bone marrow response and cytogenetics proceed to standard consolidation therapy once blood counts have recovered. Patients with M3 bone marrow status at day 28 of induction therapy are taken off the protocol. All other patients are assigned to the augmented treatment regimen.

Beginning on day 28 of induction chemotherapy, patients receive standard consolidation chemotherapy comprising VCR IV on day 0 and oral mercaptopurine (MP) on days 0-27. Patients without CNS disease at diagnosis receive MTX IT on days 7, 14, 21, and 28. Patients with CNS disease at diagnosis receive MTX IT on day 7 and cranial irradiation 5 days a week for 2 weeks. Patients with testicular disease receive bilateral testicular radiotherapy 5 days a week for 1 week and then for 3 consecutive days during the next week.

NOTE: As of 3/8/2004, patients with T-cell disease who did not achieve M1 marrow status by day 14 of induction OR who did not receive augmented induction and/or consolidation (regardless of early marrow status) receive cranial irradiation.

* Arm I: Beginning on day 28 of consolidation chemotherapy, patients receive interim maintenance I chemotherapy comprising oral DM twice daily on days 0-4 and 28-32; VCR IV on days 0 and 28; oral MTX on days 0, 7, 14, 21, 28, 35, 42, and 49; oral MP on days 0-49; and MTX IT on day 28.

Beginning on day 56 of interim maintenance I chemotherapy, patients receive delayed intensification chemotherapy comprising oral DM twice daily on days 0-6 and 14-20; VCR IV and doxorubicin (DOX) IV over 15 minutes to 2 hours on days 0, 7, and 14; PEG-ASP IM on day 3; cyclophosphamide (CTX) IV over 20-30 minutes on day 28; oral thioguanine (TG) on days 28-41; ARA-C IV or subcutaneously (SC) daily on days 28-31 and 35-38; and MTX IT on days 0 and 28.

Beginning on day 56 of delayed intensification chemotherapy, patients receive interim maintenance II chemotherapy identical to interim maintenance I chemotherapy except patients receive MTX IT on days 0 and 28.

Beginning on day 56 of interim maintenance II chemotherapy, patients receive maintenance chemotherapy comprising oral DM twice daily on days 0-4, 28-32, and 56-60; VCR IV on days 0, 28, and 56; oral MP on days 0-83; oral MTX on days 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, and 77; and MTX IT on day 0.

* Arm II: Patients receive interim maintenance I chemotherapy, delayed intensification chemotherapy, and interim maintenance II chemotherapy as in arm I. Beginning on day 56 of interim maintenance II chemotherapy, patients then receive a second course of delayed intensification chemotherapy followed by maintenance chemotherapy as in arm I.
* Arm III: Beginning on day 28 of consolidation chemotherapy, patients receive interim maintenance I chemotherapy comprising VCR IV; escalating doses of MTX IV on days 0, 10, 20, 30, and 40; and MTX IT on day 30. Patients then receive delayed intensification chemotherapy as in arm I. Patients receive interim maintenance II chemotherapy as in interim maintenance I chemotherapy, but with IV MTX starting at 2/3 of the maximum tolerated dose (MTD) attained in interim maintenance I chemotherapy. Patients then receive maintenance chemotherapy as in arm I.
* Arm IV: Patients receive interim maintenance I chemotherapy as in arm III, delayed intensification chemotherapy as in arm I, interim maintenance II chemotherapy as in arm III, delayed intensification II chemotherapy as in arm II, and maintenance chemotherapy as in arm I.
* Augmented Treatment: Patients receive induction chemotherapy comprising daunorubicin IV continuously for 48 hours beginning no later than day 21; oral DM twice daily on days 14-27; and VCR IV on days 14 and 21. Patients without CNS disease at diagnosis receive MTX IT on days 21 and 35. Patients with CNS disease at diagnosis receive MTX IT on days 21 and 28.

NOTE: Patients with T-cell disease should re-start with augmented consolidation and proceed as per the augmented regimen.

Beginning on day 35 of induction chemotherapy, patients receive consolidation therapy comprising CTX IV over 20-30 minutes on days 0 and 28; oral MP on days 0-13 and 28-41; ARA-C IV or SC daily on days 0-3, 7-10, 28-31, and 35-38; VCR IV on days 14, 21, 42, and 49; and PEG-ASP IM on days 14 and 42. Patients without CNS disease at diagnosis receive MTX IT on days 7, 14, and 21. Patients with CNS disease at diagnosis receive MTX IT on day 7 and cranial irradiation as in the randomized treatment section. Patients with testicular leukemia receive radiotherapy as in the randomized treatment section.

Beginning on day 63 of consolidation chemotherapy, patients receive interim maintenance I chemotherapy comprising VCR IV on days 0, 10, 20, 30, and 40; escalating doses of MTX IV on days 10, 20, 30, and 40; PEG-ASP IM on days 1 and 21; and MTX IT on days 0 and 30.

Beginning on day 56 of interim maintenance I chemotherapy, patients receive delayed intensification I chemotherapy comprising oral DM twice daily on days 0-6 and 14-20; VCR IV on days 0, 7, 14, 42, and 49; DOX IV over 15 minutes to 2 hours on days 0, 7, and 14; PEG-ASP IM on days 3 and 42; CTX IV over 20-30 minutes on day 28; oral TG on days 28-41; ARA-C IV or SC daily on days 28-31 and 35-38; and MTX IT on days 0 and 28.

NOTE: Patients with T-cell disease who are in interim maintenance I chemotherapy with escalating IV methotrexate should continue this phase and then proceed as per the augmented regimen. If these patients are receiving conventional interim maintenance chemotherapy with oral methotrexate, they should stop and restart the interim maintenance as per the augmented regimen. These patients receive cranial irradiation starting on day 28 of delayed intensification II chemotherapy.

Beginning on day 56 of delayed intensification I chemotherapy, patients receive interim maintenance II chemotherapy as in interim maintenance I chemotherapy, but with IV MTX starting at 2/3 of the MTD attained in interim maintenance I chemotherapy.

NOTE: Patients with T-cell disease who are in delayed intensification I chemotherapy proceed with this phase, with the addition of 2 vincristine doses on days 42 and 49 and PEG-ASP on day 42. These patients then proceed as per the augmented regimen with the addition of cranial irradiation starting on day 28 of delayed intensification II chemotherapy.

NOTE: Patients with T-cell disease who are within 4 months of completing delayed intensification I chemotherapy and have not received interim maintenance II chemotherapy with escalating IV methotrexate or delayed intensification II chemotherapy receive a course of interim maintenance chemotherapy and delayed intensification II chemotherapy according to the augmented regimen. If these patients have received interim maintenance II chemotherapy with escalating IV methotrexate, they receive delayed intensification II chemotherapy according to the augmented regimen. These patients also receive cranial irradiation starting on day 28 of delayed intensification II chemotherapy and then proceed to maintenance therapy.

Beginning on day 56 of interim maintenance II chemotherapy, patients receive delayed intensification II chemotherapy as in delayed intensification I chemotherapy.

Beginning on day 56 of delayed intensification II chemotherapy, patients receive maintenance chemotherapy comprising oral DM twice daily on days 0-4, 28-32, and 56-60; VCR IV on days 0, 28, and 56; oral MP on days 0-83; oral MTX on days 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, and 77; and MTX IT on day 0.

Patients are followed every 4-8 weeks for one year, every 3 months for one year, every 6 months for one year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 2,037 randomized patients will be accrued for this study within 3.75 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of previously untreated B-cell precursor acute lymphoblastic leukemia

  * More than 25% L1 or L2 lymphoblasts
  * No more than 25% L3 lymphoblasts
  * WBC < 50,000/mm^3
* No T-cell precursor acute lymphoblastic leukemia by immunophenotyping
* Massive lymphadenopathy, massive splenomegaly, or large mediastinal mass allowed
* CNS or testicular leukemia allowed
* No patients found to have t(8;14)(q24;q32), t(8;22)(q24;q11), and t(2;8)(p11-p12;q24) (characteristic of Burkitt's lymphoma)

PATIENT CHARACTERISTICS:

Age:

* 1 to 9

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No more than 72 hours since prior intrathecal cytarabine

Endocrine therapy:

* At least 30 days since prior systemic corticosteroids given for more than 48 hours
* Prior corticosteroids for mediastinal mass causing superior mediastinal syndrome allowed
* Prior or concurrent inhaled corticosteroids allowed

Radiotherapy:

* Prior radiotherapy for mediastinal mass causing superior mediastinal syndrome allowed
* No concurrent spinal radiotherapy

Surgery:

* Not specified

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3054 (Actual)
Dates: Start 2000-06; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | Time of randomization
  The primary outcome index used in examining the randomized treatment groups will be event free survival (EFS) from the time of randomization (i.e., end of Consolidation), where the life table events will consist of the first occurrence of leukemic relapse at any site, death, or occurrence of a second malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Yousif H. Matloub, MD, Study Chair — University of Wisconsin, Madison
Locations (130):
- United States (116):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - General Robert Huyser Cancer Center at David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Mountain States Tumor Institute - Boise, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis/St. Paul, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Valerie Fund Children's Center at Atlantic Health, Summit, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Comprehensive Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Dakota Cancer Institute at Innovis Health - Dakota Clinic, Fargo, North Dakota
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Doernbecher Children's Hospital at Oregon Health & Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - MD Anderson Cancer Center at University of Texas, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - Methodist Cancer Center at Methodist Specialty and Transplant Hospital, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Cabell Huntington Hospital, Huntington, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Australia (3):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (7):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Western Ontario, London, Ontario
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Starship Children's Health, Auckland, New Zealand
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Background] Bruggers CS, Moyer-Mileur LJ, Ransdall L: Body composition, bone mineral acquisition, and cardiovascular fitness in children with standard risk acute lymphoblastic leukemia: response to a home-based exercise and nutrition education program. [Abstract] 2006 Pediatric Academic Societies' Annual Meeting, April 29 - May 2, San Francisco, CA. A-3505.46, 2006.
- [Background] Matloub Y, Asselin BL, Stork LC, et al.: Outcome of children with T-Cell acute lymphoblastic leukemia (T-ALL) and standard risk (SR) features: results of CCG-1952, CCG-1991 and POG 9404. [Abstract] Blood 104 (11): A-680, 195a, 2004.
- [Background] Fernandez CV, Kodish E, Taweel S, Shurin S, Weijer C; Children's Oncology Group. Disclosure of the right of research participants to receive research results: an analysis of consent forms in the Children's Oncology Group. Cancer. 2003 Jun 1;97(11):2904-9. doi: 10.1002/cncr.11391. PMID 12767106
- [Result] Matloub Y, Bostrom BC, Hunger SP, Stork LC, Angiolillo A, Sather H, La M, Gastier-Foster JM, Heerema NA, Sailer S, Buckley PJ, Thomson B, Cole C, Nachman JB, Reaman G, Winick N, Carroll WL, Devidas M, Gaynon PS. Escalating intravenous methotrexate improves event-free survival in children with standard-risk acute lymphoblastic leukemia: a report from the Children's Oncology Group. Blood. 2011 Jul 14;118(2):243-51. doi: 10.1182/blood-2010-12-322909. Epub 2011 May 11. PMID 21562038
- [Result] Matloub Y, Bostrom BC, Angiolillo AL, et al.: Children with NCI standard risk acute lymphoblastic leukemia (ALL) and TEL-AML1 or favorable chromosome trisomies are almost certain to be cured with graduated intensity therapy: results of the CCG - 1991 study. [Abstract] Blood 114 (22): A-320, 2009.
- [Result] Matloub Y, Bostrom BC, Hunger SP, et al.: Escalating dose intravenous methotrexate without leucovorin rescue during interim maintenance is superior to oral methotrexate for children with standard risk acute lymphoblastic leukemia (SR-ALL): Children's Oncology Group study 1991. [Abstract] Blood 112 (11): A-9, 2008.
- [Result] Matloub Y, Angiolillo A, Bostrom B, et al.: Double delayed intensification (DDI) is equivalent to single DI (SDI) in children with National Cancer Institute (NCI) standard-risk acute lymphoblastic leukemia (SR-ALL) treated on Children's Cancer Group (CCG) clinical trial 1991 (CCG-1991). [Abstract] Blood 108 (11): A-146, 2006.
- [Derived] Matloub Y, Rabin KR, Ji L, Devidas M, Hitzler J, Xu X, Bostrom BC, Stork LC, Winick N, Gastier-Foster JM, Heerema NA, Stonerock E, Carroll WL, Hunger SP, Gaynon PS. Excellent long-term survival of children with Down syndrome and standard-risk ALL: a report from the Children's Oncology Group. Blood Adv. 2019 Jun 11;3(11):1647-1656. doi: 10.1182/bloodadvances.2019032094. PMID 31160295